CLINICAL TRIAL: NCT05547308
Title: Evaluation of Gamified Training for 3D Printed Myoelectric Prosthetic Devices in Children With Upper Congenital Limb Deficiency
Brief Title: Evaluation of 3D Printed Myoelectric Prosthetic Devices in Children With Upper Congenital Limb Deficiency
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Orlando Health, Inc. (Other)
Collaborators: Limbitless Solutions (Unknown); University of Central Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017710limbitlessprosthetic
Record Dates: First submitted 2022-04-25; First posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Limb Deformities, Congenital; Upper Extremity Deformities, Congenital; Congenital Abnormalities
MeSH Terms: conditions — Limb Deformities, Congenital; Upper Extremity Deformities, Congenital; Congenital Abnormalities

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Prosthetic device (Experimental): All subjects will receive the 3D myoelectric prosthetic device
  Interventions: Device: 3D myoelectric prosthetic device

INTERVENTIONS:
Device: 3D myoelectric prosthetic device — All subjects will use the 3D Prosthetic device and complete a variety of quality of life questionnaires.

SUMMARY:
This will be a prospective study over a 14-month duration with clinical evaluations throughout. Limitless Solutions will provide prosthetics and training system for study subjects that qualify for enrollment.

DETAILED DESCRIPTION:
Prosthetics for children are costly and those families who do get them often find that children don't use them for very long for a variety of reasons, including weight and ease of use. Limitless Solutions has developed technology to create personalized bionics for people with disabilities at an affordable cost. This will be a prospective study over a 14-month duration with clinical evaluations throughout. Limitless Solutions will provide prosthetics and training system for study subjects free of charge. During each visit, the study team will include an occupational therapist, a prosthetist, a study coordinator, and a research volunteer along with Limitless support staff and a supervising physician. Subject will complete quality of life questionnaires throughout their participation.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 7 to 17
* Congenital/infant upper limb deficiency specifically transhumeral and transradial limb deficiency as identified by Limbitless Solutions.

Exclusion Criteria:

* Non-English-speaking children and families.
* Any shoulder or wrist disarticulation will be excluded.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Quality of life and function ability will be measured through questionnaire, surveys and motor testing while using the 3D myoelectric device. | baseline thru 14 months post baseline.
  This data will be compared across the population using validated testing tools.

SECONDARY OUTCOMES:
In-person testing of motor skills by an occupational therapist using blocks and a box. | baseline thru 14 months post baseline
  Box and Blocks Test measures gross motor dexterity skills with an experienced occupational therapist with both dominant and non-dominant hand by moving blocks into a box in a specific timeframe while using the 3D myoelectric prosthetic device. This will be done at delivery of device, 5 months and 14 months after delivery.

OTHER OUTCOMES:
Children's Hand-use Experience Questionnaire | baseline thru 14 months post baseline
  Children's Hand-use Experience Questionnaire is in PDF format We have developed the questionnaire to evaluate the experience of children and adolescents in using the affected hand or hand prostheses in activities where usually two hands are needed.
PedsQL TM (Pediatric Quality of Life Inventory TM) | baseline thru 14 months post baseline
  The PedsQL Measurement Model is a questionnaire that is designed to measure health-related quality of life in healthy children and adolescents and those with acute and chronic health conditions.
The use of the GUESS system for video gaming using the myoelectric device. | baseline thru 14 months post baseline
  The GUESS is a psychometrically validated and comprehensive gaming scale with nine subscales (e.g., Usability/Playability, Creative Freedom, and Social Connectivity) and 55 items in total. The GUESS is intended for any playtesting and game evaluation purposes.
The Pediatric Outcome Data Collection Instrument is a survey | baseline thru 14 months post baseline
  The Pediatric Outcomes Data Collection Instrument (PODCI) is an outcomes assessment tool developed to allow measurement of health-related quality of life in children with disorders having musculoskeletal impact. This can be patient or parent reported and addresses activities of daily living.
Psychosocial questionnaire to be completed by both patient and parent | 14 month post baseline
  This survey is designed to qualitatively identify any influence the use of the prosthetic device has throughout the study and for qualitative comparison across the patient population.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Manero, PhD, Study Director — Limbitless Solutions
Locations (1):
- Orlando Health Arnold Palmer Hospital for Children, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Blough DK, Hubbard S, McFarland LV, Smith DG, Gambel JM, Reiber GE. Prosthetic cost projections for servicemembers with major limb loss from Vietnam and OIF/OEF. J Rehabil Res Dev. 2010;47(4):387-402. doi: 10.1682/jrrd.2009.04.0037. PMID 20803406
- [Result] Canfield MA, Honein MA, Yuskiv N, Xing J, Mai CT, Collins JS, Devine O, Petrini J, Ramadhani TA, Hobbs CA, Kirby RS. National estimates and race/ethnic-specific variation of selected birth defects in the United States, 1999-2001. Birth Defects Res A Clin Mol Teratol. 2006 Nov;76(11):747-56. doi: 10.1002/bdra.20294. PMID 17051527
- See also: Limbitless Solutions, Inc. — http://limbitless-solutions.org/about-us/